CLINICAL TRIAL: NCT01758328
Title: A Phase I Dose Escalation Trial of WT1-specific Donor-derived T Cells Following T-Cell Depleted Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Dose Escalation Trial of WT1-specific Donor-derived T Cells Following T-Cell Depleted Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-175
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: BUSULFAN; FLUDARABINE; G-CSF; MELPHALAN; RABBIT ATG WT1; PEPTIDE SPECIFIC T CELLS; 12-175
MeSH Terms: conditions — Multiple Myeloma | interventions — Busulfan; Melphalan; fludarabine; Antilymphocyte Serum

ARMS (1):
- Pts with Mutiple myeloma (Experimental): Patients will undergo a preparative regimen with busulfan, melphalan, fludarabine, and anti-thymocyte globulin (ATG), and a T cell depleted stem cell transplant from a histocompatible related or unrelated donor. Hematopoietic stem cell donors for this trial will include individuals who are 10/10 HLA matched or one antigen or allele mismatched at the HLA-A, B, C, DRB1 or DQB1 locus, as defined by high resolution methods .Donors who are 8/10 HLA matched with an antigen or allele mismatched at HLA-DQB1 and at one other locus will also be eligible for the trial. The administration of WT1-specific cytotoxic T cells (WT1 CTLs) post transplantation is integrated to induce complete remissions in patients with residual disease and to decrease the rate of relapse following the allogeneic transplant.
  Interventions: Drug: busulfan; Drug: melphalan; Drug: fludarabine; Biological: anti-thymocyte globulin (ATG); Procedure: a T cell depleted stem cell transplant

INTERVENTIONS:
Drug: busulfan
Drug: melphalan
Drug: fludarabine
Biological: anti-thymocyte globulin (ATG)
Procedure: a T cell depleted stem cell transplant

SUMMARY:
The purpose of this study is to test the safety of specialized white cells from the donor at different doses. They are called WT1 sensitized T cells. They have been grown in the lab and are immunized against a protein. The protein is called the Wilms' tumor protein, or WT1. The multiple myeloma cells make and express this protein". The investigators want to learn whether the WT1 sensitized T cells will attach to the protein and kill the myeloma cells. The investigators want to find out what effects, good and/or bad, it has on the patient and multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis:

* Patient must have multiple myeloma that has either relapsed or remains refractory following autologous stem cell transplantation and patients who have plasma cell leukemia at diagnosis.
* Patients with relapsed multiple myeloma following autologous stem cell transplantation who achieved < partial response following additional chemotherapy or who achieved < PR at 3 months following autologous stem cell transplantation and patients with plasma cell leukemia at diagnosis.

DONOR: Patients must have a healthy HLA matched or mismatched related or unrelated donor who is willing to receive G-CSF injections and undergo apheresis for PBSC collection, or undergo a marrow harvesting procedure.

* HLA-matched related and unrelated donors Patients who have an HLA-matched related or unrelated donor are eligible for entry on this protocol. This will include a healthy donor who is genotypically matched at all A, B, C, DRB1 and DQB1 loci, as tested by DNA analysis.
* HLA- mismatched related and unrelated donors
* Patients who do not have an HLA-matched donor but have a related or unrelated donor who have one antigen or one allele mismatch at the HLA A, B, C, DRB1 or DQB1 loci or who have two mismatches, at HLA-DQB1 and at one other locus, will be eligible for entry on this protocol.

The following inclusion criteria are also required:

* Patients should be ≥ 21, < 73 years old.
* Patients may be of either gender or any ethnic background.
* Patients must have a Karnofsky (adult) or Performance Status > 70%
* Patients must have adequate organ function measured by:

  1. Cardiac: asymptomatic or if symptomatic then LVEF at rest must be > 50% and must improve with exercise.
  2. Hepatic: < 3x ULN ALT and < 1.5 total serum bilirubin, unless there is congenital benign hyperbilirubinemia.
  3. Renal: serum creatinine <1.2 mg/dl or if serum creatinine is outside the normal range, then CrCl > 40 ml/min (measured or calculated/estimated) with dose adjustment of Fludarabine for <70ml/min.
  4. Pulmonary: asymptomatic or if symptomatic, DLCO > 50% of predicted (corrected for hemoglobin)
* Each patient must be willing to participate as a research subject and must sign an informed consent form.

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Active viral, bacterial or fungal infection
* Patient seropositive for HIV-I/II; HTLV -I/II
* Patients who have had a previous malignancy that is not in remission.
* Patients with known hypersensitivity to mouse proteins (murine antibodies in ISOLEX) if receiving SBA-E- bone marrow, or chicken egg products.

Ages: 21 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
assess the toxicities | 21 days
  DLT will be defined as a grade III or greater toxicity developing within 3 weeks of the T cell infusion, as graded by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4 or new development of grade II-IV acute GVHD within 3 weeks of the T cell infusion that requires treatment with systemic glucocorticosteroids. Patients will be evaluated for 21 days for grade III or greater toxicities.
maximum tolerated dose (MTD) | 1 year
  Patients will also be monitored for secondary or immune-mediated graft rejection and or onset of grade II-IV acute GVHD following the administration of WT1-specific T-cell infusions. Because patients may still have transplantation associated cytopenia or may have residual disease that may be associated with cytopenias, hematologic toxicity will be excluded in assessing DLT. All patients will be observed for a minimum of 3 weeks after the first WT-1 peptide sensitized T-cell infusion before the dose can be escalated.

SECONDARY OUTCOMES:
serologic response | 2 years
  In addition, patients will be monitored for serologic responses of their myelomas. The time at which the response was achieved will be recorded for all patients and summarized by dose level. The data derived from these studies will provide an initial assessment of the effects of the T cell infusions.
survival | 2 years
  To quantitate the number of WT1-specific T cells in the blood and marrow at defined intervals post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Giralt, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/